CLINICAL TRIAL: NCT02010255
Title: A Phase 2, Multicenter, Open-Label Study to Investigate the Safety and Efficacy of Sofosbuvir/Ledipasvir Fixed-Dose Combination + Ribavirin Administered in Subjects Infected With Chronic HCV Who Have Advanced Liver Disease or Are Post-Liver Transplant
Brief Title: Ledipasvir/Sofosbuvir Fixed-Dose Combination Plus Ribavirin in Participants With Chronic HCV With Advanced Liver Disease or Post-Liver Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-0124; 2013-002802-30 (EudraCT Number)
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2016-05

CONDITIONS: Chronic HCV Infection
MeSH Terms: interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (14):
- Cohort A, Group 1 (12 wk): CPT Class B (7-9) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class B (CPT score 7-9)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort A, Group 1 (24 wk): CPT Class B (7-9) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 24 weeks in participants with CPT Class B (CPT score 7-9)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort A, Group 2 (12 wk): CPT Class C (10-12) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class C (CPT score 10-12)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort A, Group 2 (24 wk): CPT Class C (10-12) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 24 weeks in participants with CPT Class C (CPT score 10-12)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 3 (12 wk): F0-F3 Fibrosis (Experimental): LDV/SOF (90/400 mg) plus RBV (weight-based: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with Fibrosis Stage F0-F3
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 3 (24 wk): F0-F3 Fibrosis (Experimental): LDV/SOF (90/400 mg) plus RBV (weight-based: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 24 weeks in participants with Fibrosis Stage F0-F3
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 4 (12 wk): CPT Class A (5-6) (Experimental): LDV/SOF (90/400 mg) plus RBV (weight-based: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with CPT Class A (CPT score 5-6)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 4 (24 wk): CPT Class A (5-6) (Experimental): LDV/SOF (90/400 mg) plus RBV (weight-based: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 24 weeks in participants with CPT Class A (CPT score 5-6)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 5 (12 wk): CPT Class B (7-9) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class B (CPT score 7-9)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 5 (24 wk): CPT Class B (7-9) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 24 weeks in participants with CPT Class B (CPT score 7-9)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 6 (12 wk): CPT Class C (10-12) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class C (CPT score 10-12)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 6 (24 wk): CPT Class C (10-12) (Experimental): LDV/SOF (90/400 mg) plus RBV (starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 24 weeks in participants with CPT Class C (CPT score 10-12)
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 7 (12 wk): FCH (Experimental): LDV/SOF (90/400 mg) plus RBV (weight-based: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with FCH
  Interventions: Drug: LDV/SOF; Drug: RBV
- Cohort B, Group 7 (24 wk): FCH (Experimental): LDV/SOF (90/400 mg) plus RBV (weight-based: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 24 weeks in participants with FCH
  Interventions: Drug: LDV/SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — LDV/SOF FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: RBV — RBV tablets administered orally in a divided daily dose

SUMMARY:
This study will evaluate ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) plus ribavirin (RBV) in participants with advanced liver disease or posttransplant and chronic genotype 1 or 4 hepatitis C virus (HCV) infection.

* Cohort A: decompensated cirrhosis (advanced liver disease), no prior liver transplant;
* Cohort B: post-liver transplant, with or without cirrhosis;
* Group assignment within cohorts is based on severity of liver impairment at screening (Child-Pugh-Turcotte (CPT) score for participants with cirrhosis; fibrosis; or presence of disease for fibrosing cholestatic hepatitis (FCH) groups)
* Randomization is 1:1 within groups to 12 or 24 weeks of LDV/SOF+RBV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Chronic genotype 1 and/or 4 HCV infection
* Normal ECG
* Negative serum pregnancy test for female subjects
* Male subjects and female subjects of childbearing potential must agree to use contraception
* Able to comply with the dosing instructions for study drug and able to complete the study schedule of assessments, including all required post treatment visits

Exclusion Criteria:

* Serious or active medical or psychiatric illness
* HIV or hepatitis B viral (HBV) infection
* Stomach disorder that could interfere with the absorption of the study drug
* Treated with an anti-HCV medication in the last 30 days
* Any prior exposure to an HCV nonstructural protein (NS)5a-specific inhibitor
* Use of human granulocyte-macrophage colony-stimulating factor (GM-CSF), epoetin alfa or other therapeutic hematopoietic agents within 2 weeks of screening
* History of clinically significant medical condition associated with other chronic liver disease
* Active spontaneous bacterial peritonitis at screening
* Females who are breastfeeding
* Infection requiring systemic antibiotics
* Participated in a clinical study with an investigational drug or biologic within the last 30 days
* Active or history (last 6 months) of drug or alcohol abuse
* History of organ transplant other than liver, kidney, or corneal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shampa De-Oertel, PhD, Study Director — Gilead Sciences
Locations (34):
- Australia (2):
  - Royal Prince Alfred Hospital, University of Sydney, Camperdown, New South Wales
  - Austin Repatriation Hospital (Melbourne) // Victorian Transplant Centre, Heidelberg, Victoria
- Austria (2):
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Medizinische Universitat Wien, Vienna
- Belgium (2):
  - UCL St-Luc Brussels, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Canada (6):
  - Division of Gastroenterology, University of Alberta, Edmonton, Edmonton, Alberta
  - University of British Columbia and Vancouver General Hospital, Vancouver, British Columbia
  - London Health Sciences Centre-University Hospital, London, Ontario
  - University Health Network // Toronto General Hospital, Toronto, Ontario
  - Hopital St. Luc, Montreal, Quebec
  - McGill University Health Centre \ Royal Victoria Hospital, Montreal, Quebec
- France (4):
  - Hospital Beaujon, Clichy
  - Hospital Mondor \ Service d'Hépatologie et de Gastroentérologie,, Créteil
  - Hopital Saint-Eloi, Montpellier
  - Hopital Paul Brousse, Villejuif
- Germany (4):
  - Universitätsklinikum RWTH Aachen, Aachen
  - Universitätsklinikum Essen - klinikum für Gastroenterolgie und Hepatologie, Essen
  - University Hospital Johann Wolfgang Goethe University, Department of Internal Medicine I, Frankfurt
  - Medical School of Hannover, Hanover
- Italy (2):
  - IRCCS Cà Grande Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera San Giovanni, Battista di Torino \ Professor of Gastroenterology-San Giovanni Battista Hospital-University of Torino, Torino
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus MC in Rotterdam, Rotterdam
- Auckland City Hospital, Auckland, New Zealand
- Spain (4):
  - Hospital General Universitari Vall d' Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Puerta de Hierro, Madrid, Madrid
  - Hospital Universitario y Politecnico La Fe de Valencia, Valencia
- Switzerland (2):
  - University of Berne, Bern
  - University Hospital Zurich, Zurich
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Infirmary of Edinburgh \ Scottish Liver Transplant Unit-Edinburgh, Edinburgh
  - Kings College Hospital, Institute of Liver Studies, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Manns M, Samuel D, Gane EJ, Mutimer D, McCaughan G, Buti M, Prieto M, Calleja JL, Peck-Radosavljevic M, Mullhaupt B, Agarwal K, Angus P, Yoshida EM, Colombo M, Rizzetto M, Dvory-Sobol H, Denning J, Arterburn S, Pang PS, Brainard D, McHutchison JG, Dufour JF, Van Vlierberghe H, van Hoek B, Forns X; SOLAR-2 investigators. Ledipasvir and sofosbuvir plus ribavirin in patients with genotype 1 or 4 hepatitis C virus infection and advanced liver disease: a multicentre, open-label, randomised, phase 2 trial. Lancet Infect Dis. 2016 Jun;16(6):685-697. doi: 10.1016/S1473-3099(16)00052-9. Epub 2016 Feb 18. PMID 26907736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe, Canada, Australia, and New Zealand. The first participant was screened on 14 January 2014. The last study visit occurred on 27 August 2015.
Pre-assignment Details: * Cohort A: decompensated cirrhosis [advanced liver disease], no prior liver transplant;
  * Cohort B: post-liver transplant, with or without cirrhosis;
  * Group assignment within cohorts was based on severity of liver impairment at screening [or presence of disease for FCH groups];
  * Randomization was 1:1 within groups to 12 or 24 weeks of treatment.
Groups:
- Cohort A, Group 1 (12 wk): CPT Class B (7-9): Ledipasvir/sofosbuvir (Harvoni®; LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet once daily plus ribavirin (RBV) tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with Child-Pugh-Turcotte (CPT) Class B (CPT score 7-9).
  CPT scores grade the severity of cirrhosis and are used to determine the need for liver transplantation. Scores can range from 5 to 15 (maximum score for study was 12); higher scores indicate greater severity of disease.
- Cohort A, Group 1 (24 wk): CPT Class B (7-9); Cohort B, Group 5 (24 wk): CPT Class B (7-9): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 24 weeks in participants with CPT Class B (CPT score 7-9).
- Cohort A, Group 2 (12 wk): CPT Class C (10-12); Cohort B, Group 6 (12 wk): CPT Class C (10-12): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class C (CPT score 10-12).
- Cohort A, Group 2 (24 wk): CPT Class C (10-12); Cohort B, Group 6 (24 wk): CPT Class C (10-12): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 24 weeks in participants with CPT Class C (CPT score 10-12).
- Cohort B, Group 3 (12 wk): F0-F3 Fibrosis: LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with Fibrosis Stage F0-F3.
  F0: no fibrosis; F1: portal fibrosis without septa; F2: portal fibrosis with rare septa, F3: numerous septa without cirrhosis; F4: cirrhosis.
- Cohort B, Group 3 (24 wk): F0-F3 Fibrosis: LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 24 weeks in participants with Fibrosis Stage F0-F3.
- Cohort B, Group 4 (12 wk): CPT Class A (5-6): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with CPT Class A (CPT score 5-6).
- Cohort B, Group 4 (24 wk): CPT Class A (5-6): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 24 weeks in participants with CPT Class A (CPT score 5-6).
- Cohort B, Group 5 (12 wk): CPT Class B (7-9): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class B (CPT score 7-9).
- Cohort B, Group 7 (12 wk): FCH: LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with FCH
- Cohort B, Group 7 (24 wk): FCH: LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 24 weeks in participants with FCH
Period: Overall Study
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Started | 28 | 28 | 25 | 26 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 5 | 3 | 3
Completed | 22 | 26 | 18 | 20 | 48 | 49 | 33 | 32 | 21 | 23 | 1 | 4 | 3 | 2
Not Completed | 6 | 2 | 7 | 6 | 4 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 1
Not completed — Death | 0 | 1 | 4 | 4 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 4 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrew Consent | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but Not Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled and received at least one dose of study drug
Groups:
- Cohort A, Group 1 (12 wk): CPT Class B (7-9); Cohort B, Group 5 (12 wk): CPT Class B (7-9): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class B (CPT score 7-9).
- Cohort B, Group 3 (12 wk): F0-F3 Fibrosis: LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (weight-based divided daily dose: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg) for 12 weeks in participants with Fibrosis Stage F0-F3.
- Total: Total of all reporting groups
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH | Total
Number analyzed (Participants) | 28 | 28 | 25 | 26 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 5 | 3 | 2 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (9.9) | 56 (8.6) | 58 (8.1) | 54 (10.7) | 58 (7.9) | 59 (6.9) | 57 (7.2) | 62 (7.5) | 58 (8.0) | 60 (10.2) | 62 (4.6) | 62 (9.2) | 58 (2.6) | 56 (2.8) | 58 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 10 | 6 | 11 | 10 | 6 | 7 | 7 | 8 | 1 | 0 | 1 | 1 | 82
  Male | 23 | 19 | 15 | 20 | 41 | 39 | 28 | 26 | 15 | 15 | 2 | 5 | 2 | 1 | 251
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 3 | 8 | 4 | 8 | 5 | 7 | 3 | 4 | 1 | 2 | 0 | 0 | 57
  Not Hispanic or Latino | 22 | 22 | 22 | 18 | 48 | 41 | 29 | 26 | 19 | 19 | 2 | 3 | 3 | 2 | 276
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5
  White | 25 | 28 | 23 | 25 | 50 | 47 | 33 | 30 | 21 | 21 | 3 | 5 | 2 | 1 | 314
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 1 | 7
  Native Hawaiian or Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Other | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 0 | 1 | 3 | 2 | 0 | 2 | 2 | 2 | 1 | 0 | 0 | 2 | 0 | 16
  Canada | 6 | 5 | 4 | 1 | 8 | 6 | 4 | 5 | 4 | 5 | 0 | 0 | 0 | 1 | 49
  Austria | 2 | 2 | 1 | 0 | 8 | 2 | 2 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 23
  Netherlands | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 8
  Belgium | 1 | 2 | 3 | 0 | 3 | 3 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 16
  Italy | 2 | 1 | 2 | 1 | 2 | 2 | 3 | 1 | 3 | 3 | 1 | 2 | 0 | 0 | 23
  United Kingdom | 5 | 3 | 0 | 1 | 8 | 9 | 4 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 36
  Australia | 1 | 1 | 7 | 4 | 0 | 2 | 3 | 3 | 2 | 2 | 0 | 1 | 0 | 1 | 27
  France | 1 | 1 | 1 | 4 | 4 | 5 | 6 | 3 | 3 | 3 | 0 | 0 | 1 | 0 | 32
  Switzerland | 1 | 4 | 1 | 2 | 4 | 3 | 4 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 23
  Germany | 2 | 4 | 3 | 3 | 6 | 5 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 28
  Spain | 6 | 5 | 2 | 7 | 4 | 8 | 5 | 5 | 3 | 4 | 1 | 2 | 0 | 0 | 52
Hepatitis C Virus (HCV) RNA [Mean (Standard Deviation); unit: log 10 IU/mL] | 6.0 (0.49) | 5.9 (0.56) | 5.6 (0.58) | 5.7 (0.44) | 6.4 (0.72) | 6.5 (0.44) | 6.3 (0.58) | 6.5 (0.55) | 6.1 (0.78) | 6.2 (0.85) | 6.0 (0.49) | 6.5 (0.50) | 7.3 (0.72) | 6.0 (0.41) | 6.2 (0.66)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 11 | 14 | 16 | 17 | 12 | 5 | 9 | 5 | 5 | 9 | 2 | 0 | 0 | 1 | 106
  ≥ 800,000 IU/mL | 17 | 14 | 9 | 9 | 40 | 44 | 25 | 28 | 17 | 14 | 1 | 5 | 3 | 1 | 227
HCV Genotype [Number; unit: participants]
  Genotype 1a | 13 | 12 | 13 | 12 | 27 | 29 | 14 | 13 | 11 | 13 | 1 | 1 | 2 | 2 | 163
  Genotype 1b | 12 | 13 | 11 | 11 | 18 | 15 | 16 | 15 | 9 | 7 | 1 | 4 | 1 | 0 | 133
  Genotype 4 | 3 | 3 | 1 | 3 | 7 | 5 | 4 | 5 | 2 | 3 | 1 | 0 | 0 | 0 | 37
IL28b Status [Number; unit: participants]
  CC | 6 | 9 | 7 | 4 | 9 | 10 | 3 | 7 | 3 | 5 | 0 | 3 | 0 | 1 | 67
  CT | 18 | 10 | 10 | 15 | 31 | 25 | 23 | 21 | 12 | 11 | 2 | 2 | 3 | 1 | 184
  TT | 4 | 9 | 8 | 7 | 12 | 14 | 8 | 5 | 7 | 7 | 1 | 0 | 0 | 0 | 82

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were randomized and received at least one dose of study drug. Participants in Cohort A who received a liver transplant prior to the lower bound of the Posttreatment Week 12 visit were not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 25 | 21 | 25 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 5 | 3 | 2
percentage of participants | 84.6 | 96.0 | 81.0 | 76.0 | 94.2 | 100.0 | 97.1 | 97.0 | 95.5 | 100.0 | 33.3 | 80.0 | 100.0 | 100.0

2. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set: participants who were randomized and received at least one dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 28 | 28 | 25 | 26 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 5 | 3 | 2
percentage of participants
  Discontinued LDV/SOF | 3.6 | 3.6 | 0.0 | 7.7 | 1.9 | 0.0 | 0.0 | 3.0 | 0.0 | 0.0 | 0.0 | 20.0 | 0.0 | 0.0
  Discontinued Any Study Drug | 3.6 | 7.1 | 16.0 | 23.1 | 5.8 | 6.1 | 0.0 | 15.2 | 18.2 | 17.4 | 33.3 | 20.0 | 0.0 | 0.0

3. Secondary Outcome: Percentage of Participants With SVR 2 Weeks After Discontinuation of Therapy (SVR2)
Description: SVR2 was defined as HCV RNA < LLOQ at 2 weeks after stopping study treatment.
Time Frame: Posttreatment Week 2
Population: Full Analysis Set. Participants in Cohort A who received a liver transplant prior to the lower bound of the Posttreatment Week 2 visit were not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 26 | 23 | 25 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 5 | 3 | 2
percentage of participants | 96.2 | 100.0 | 91.3 | 80.0 | 98.1 | 100.0 | 100.0 | 97.0 | 95.5 | 100.0 | 100.0 | 80.0 | 100.0 | 100.0

4. Secondary Outcome: Percentage of Participants With SVR 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set. Participants in Cohort A who received a liver transplant prior to the lower bound of the Posttreatment Week 4 visit were not included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 26 | 22 | 25 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 5 | 3 | 2
Percentage of participants | 88.5 | 100.0 | 90.9 | 80.0 | 94.2 | 100.0 | 97.1 | 97.0 | 95.5 | 100.0 | 100.0 | 80.0 | 100.0 | 100.0

5. Secondary Outcome: Percentage of Participants With SVR 8 Weeks After Discontinuation of Therapy (SVR8)
Description: SVR8 was defined as HCV RNA < LLOQ at 8 weeks after stopping study treatment.
Time Frame: Posttreatment Week 8
Population: Full Analysis Set. Participants in Cohort A who received a liver transplant prior to the lower bound of the Posttreatment Week 8 visit were not included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 26 | 22 | 25 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 5 | 3 | 2
Percentage of participants | 84.6 | 96.2 | 81.8 | 80.0 | 94.2 | 100.0 | 97.1 | 97.0 | 95.5 | 100.0 | 33.3 | 80.0 | 100.0 | 100.0

6. Secondary Outcome: Percentage of Participants With SVR 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Full Analysis Set. Participants in Cohort A and 1 participant in Cohort B who received a liver transplant prior to the lower bound of the Posttreatment Week 24 visit were not included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 25 | 25 | 20 | 25 | 52 | 49 | 34 | 33 | 22 | 22 | 3 | 5 | 3 | 2
Percentage of participants | 84.0 | 96.0 | 80.0 | 76.0 | 94.2 | 100.0 | 97.1 | 97.0 | 95.5 | 100.0 | 33.3 | 80.0 | 100.0 | 100.0

7. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ on 2 consecutive measurements while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set. Participants were excluded from the analysis if they received a liver transplant while on study (with HCV RNA <LLOQ at transplant) prior to lower bound of Posttreatment Week 12 visit window.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 25 | 21 | 25 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 5 | 3 | 2
Percentage of participants | 15.4 | 4.0 | 9.5 | 4.0 | 1.9 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 33.3 | 0.0 | 0.0 | 0.0

8. Secondary Outcome: Percentage of Participants With Posttransplant Virologic Response (pTVR) at Posttransplant Week 12
Description: pTVR was defined as HCV RNA < LLOQ at Week 12 after transplant.
Time Frame: Posttreatment Week 12
Population: Participants who had a liver transplant while on study were analyzed if their last observed HCV RNA measurement prior to transplant was < LLOQ. Participants who received a transplant from an HCV-infected donor were excluded from analysis.
Measure: Number; unit: Percentage of participants
Groups:
- All LDV/SOF+RBV: All participants in the analysis are presented in a single group, regardless of randomization group assignment.
Arm/Group | All LDV/SOF+RBV
Number analyzed (Participants) | 10
Percentage of participants | 100.0

9. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 1
Time Frame: Week 1
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 27 | 25 | 26 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 5 | 3 | 2
Percentage of participants | 3.8 | 3.7 | 12.0 | 3.8 | 9.6 | 6.1 | 5.9 | 3.0 | 0.0 | 8.7 | 0.0 | 0.0 | 0.0 | 0.0

10. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 2
Time Frame: Week 2
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 27 | 25 | 26 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 5 | 3 | 2
Percentage of participants | 26.9 | 37.0 | 40.0 | 38.5 | 48.1 | 44.9 | 26.5 | 21.2 | 31.8 | 30.4 | 0.0 | 0.0 | 33.3 | 0.0

11. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 4
Time Frame: Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 27 | 25 | 26 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 4 | 3 | 2
Percentage of participants | 76.9 | 81.5 | 80.0 | 84.6 | 84.6 | 91.8 | 67.6 | 81.8 | 72.7 | 82.6 | 100 | 25 | 100.0 | 100.0

12. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 6
Time Frame: Week 6
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 27 | 24 | 25 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 4 | 3 | 2
Percentage of participants | 100.0 | 100.0 | 91.7 | 100.0 | 98.1 | 100.0 | 100.0 | 97.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

13. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 8
Time Frame: Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 27 | 24 | 25 | 52 | 49 | 34 | 32 | 22 | 23 | 3 | 4 | 3 | 2
Percentage of participants | 100.0 | 100.0 | 100.0 | 96.0 | 100.0 | 100.0 | 100.0 | 96.9 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

14. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 12
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 27 | 24 | 24 | 51 | 49 | 34 | 32 | 22 | 23 | 3 | 4 | 3 | 2
Percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 95.5 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

15. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 16
Time Frame: Week 16
Population: Participants in the Full Analysis Set who were randomized to a 24-week treatment group and had available data were analyzed. 12-week treatment groups (did not collect data past Week 12) are not presented in this table.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 22 | 49 | 32 | 23 | 4 | 2
Percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

16. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 20
Time Frame: Week 20
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 21 | 49 | 32 | 23 | 4 | 2
Percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

17. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 24
Time Frame: Week 24
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 25 | 21 | 49 | 32 | 23 | 4 | 2
Percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

18. Secondary Outcome: HCV RNA Levels and Change From Baseline at Week 1
Time Frame: Baseline; Week 1
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 27 | 24 | 25 | 52 | 49 | 34 | 33 | 22 | 23 | 3 | 5 | 3 | 2
log10 IU/mL
  Week 1 | 2.44 (0.665) | 2.47 (0.696) | 2.32 (0.868) | 2.50 (0.645) | 2.38 (0.716) | 2.38 (0.653) | 2.64 (0.784) | 2.81 (0.729) | 2.63 (0.780) | 2.75 (0.888) | 2.97 (0.229) | 3.73 (0.434) | 2.91 (0.825) | 2.28 (0.620)
  Change at Week 1 | -3.60 (0.535) | -3.39 (0.634) | -3.28 (0.735) | -3.20 (0.610) | -3.98 (0.611) | -4.12 (0.538) | -3.70 (0.489) | -3.65 (0.562) | -3.50 (0.666) | -3.44 (0.789) | -3.06 (0.645) | -2.74 (0.446) | -4.40 (0.503) | -3.76 (0.213)

19. Secondary Outcome: HCV RNA Levels and Change From Baseline at Week 2
Time Frame: Baseline; Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 27 | 25 | 26 | 52 | 48 | 33 | 33 | 22 | 23 | 3 | 5 | 3 | 2
log10 IU/mL
  Week 2 | 1.76 (0.668) | 1.70 (0.579) | 1.71 (0.625) | 1.72 (0.573) | 1.62 (0.604) | 1.49 (0.477) | 1.92 (0.839) | 1.97 (0.607) | 1.86 (0.607) | 2.00 (0.718) | 2.08 (0.378) | 2.81 (0.709) | 1.85 (0.731) | 1.65 (0.122)
  Change at Week 2 | -4.29 (0.534) | -4.17 (0.538) | -3.92 (0.610) | -3.99 (0.566) | -4.74 (0.733) | -5.00 (0.522) | -4.42 (0.729) | -4.48 (0.583) | -4.26 (0.708) | -4.20 (0.764) | -3.95 (0.796) | -3.66 (0.601) | -5.46 (0.756) | -4.38 (0.285)

20. Secondary Outcome: HCV RNA Levels and Change From Baseline at Week 4
Time Frame: Baseline; Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 27 | 24 | 25 | 52 | 49 | 34 | 32 | 22 | 23 | 3 | 4 | 3 | 2
log10 IU/mL
  Week 4 | 1.26 (0.257) | 1.20 (0.148) | 1.23 (0.205) | 1.18 (0.147) | 1.23 (0.247) | 1.18 (0.129) | 1.29 (0.301) | 1.21 (0.154) | 1.25 (0.199) | 1.32 (0.408) | 1.15 (0.000) | 1.56 (0.585) | 1.15 (0.000) | 1.15 (0.000)
  Change at Week 4 | -4.78 (0.430) | -4.66 (0.518) | -4.45 (0.521) | -4.52 (0.492) | -5.13 (0.721) | -5.32 (0.453) | -5.05 (0.526) | -5.25 (0.518) | -4.88 (0.762) | -4.87 (0.816) | -4.89 (0.490) | -4.91 (0.240) | -6.16 (0.725) | -4.89 (0.407)

21. Secondary Outcome: HCV RNA Levels and Change From Baseline at Week 6
Time Frame: Baseline; Week 6
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 27 | 23 | 25 | 51 | 49 | 34 | 32 | 22 | 23 | 3 | 4 | 3 | 2
log10 IU/mL
  Week 6 | 1.15 (0.000) | 1.15 (0.000) | 1.17 (0.102) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000)
  Change at Week 6 | -4.90 (0.487) | -4.72 (0.535) | -4.51 (0.527) | -4.56 (0.445) | -5.21 (0.728) | -5.35 (0.436) | -5.19 (0.577) | -5.31 (0.557) | -4.98 (0.779) | -5.05 (0.851) | -4.89 (0.490) | -5.33 (0.574) | -6.16 (0.725) | -4.89 (0.407)

22. Secondary Outcome: HCV RNA Levels and Change From Baseline at Week 8
Time Frame: Baseline; Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 27 | 24 | 24 | 52 | 49 | 34 | 31 | 22 | 23 | 3 | 4 | 3 | 2
log10 IU/mL
  Week 8 | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000)
  Change at Week 8 | -4.90 (0.487) | -4.72 (0.535) | -4.53 (0.534) | -4.60 (0.393) | -5.21 (0.722) | -5.35 (0.436) | -5.19 (0.577) | -5.31 (0.565) | -4.98 (0.779) | -5.05 (0.851) | -4.89 (0.490) | -5.33 (0.574) | -6.16 (0.725) | -4.89 (0.407)

23. Secondary Outcome: HCV RNA Levels and Change From Baseline at Week 12
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Number analyzed (Participants) | 26 | 27 | 24 | 24 | 51 | 49 | 34 | 32 | 21 | 23 | 3 | 4 | 3 | 2
log10 IU/mL
  Week 12 | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000)
  Change at Week 12 | -4.90 (0.487) | -4.72 (0.535) | -4.53 (0.534) | -4.60 (0.393) | -5.21 (0.729) | -5.35 (0.436) | -5.19 (0.577) | -5.30 (0.556) | -4.98 (0.798) | -5.05 (0.851) | -4.89 (0.490) | -5.33 (0.574) | -6.16 (0.725) | -4.89 (0.407)

24. Secondary Outcome: Percentage of Participants With a Decrease, No Change, or Increase Between Baseline and Posttreatment Week 4 in MELD Score
Description: Model for End-Stage Liver Disease (MELD) scores are used to assess prognosis and suitability for liver transplantation. Scores can range from 6 to 40; higher scores/increased scores indicate greater severity of disease.
Time Frame: Baseline to Posttreatment Week 4
Population: Full Analysis Set. Participants with cirrhosis were analyzed if they had measurements at both baseline and Posttreatment Week 4. Only groups with cirrhotic participants are presented.
Measure: Number; unit: percentage of participants
Groups:
- Cohort A, Group 1 (12 wk): CPT Class B (7-9): LDV/SOF (90/400 mg) FDC tablet once daily plus RBV tablets (divided daily dose starting at 600 mg, then adjusted ± based on tolerability [weight-based maximum: < 75 kg = 1000 mg, ≥ 75 kg = 1200 mg]) for 12 weeks in participants with CPT Class B (CPT score 7-9).
  CPT scores grade the severity of cirrhosis and are used to determine the need for liver transplantation. Scores can range from 5 to 15 (maximum score for study was 12); higher scores indicate greater severity of disease.
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12)
Number analyzed (Participants) | 24 | 22 | 21 | 20 | 32 | 32 | 21 | 23 | 2 | 4
percentage of participants
  Decrease | 70.8 | 77.3 | 81.0 | 70.0 | 28.1 | 62.5 | 66.7 | 65.2 | 50.0 | 75.0
  No Change | 12.5 | 9.1 | 14.3 | 5.0 | 31.3 | 18.8 | 14.3 | 17.4 | 50.0 | 0.0
  Increase | 16.7 | 13.6 | 4.8 | 25.0 | 40.6 | 18.8 | 19.0 | 17.4 | 0.0 | 25.0

25. Secondary Outcome: Percentage of Participants With a Decrease, No Change, or Increase Between Baseline and Posttreatment Week 4 in CPT Score
Description: CPT scores grade the severity of cirrhosis and are used to determine the need for liver transplantation. Scores can range from 5 to 15 (maximum score for entry into the study was 12); higher scores/increased scores indicate greater severity of disease. Groups are arranged by cohort, then by duration of treatment, then by CPT class at baseline.
Time Frame: Baseline to Posttreatment Week 4
Population: Full Analysis Set. Cirrhotic participants were analyzed if they had measurements at both baseline and Posttreatment Week 4. Only groups with cirrhotic participants are presented.
Measure: Number; unit: percentage of participants
Groups:
- Cohort A: Baseline CPT Class B (12 wk): Includes participants in Cohort A (12 wk) with CPT score B at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort A: Baseline CPT Class B (24 wk): Includes participants in Cohort A (24 wk) with CPT score B at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort A: Baseline CPT Class C (12 wk): Includes participants in Cohort A (12 wk) with CPT score C at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort A: Baseline CPT Class C (24 wk): Includes participants in Cohort A (24 wk) with CPT score C at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort B: Baseline CPT Class A (12 wk): Includes participants in Cohort B (12 wk) with CPT score A at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort B: Baseline CPT Class A (24 wk): Includes participants in Cohort B (24 wk) with CPT score A at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort B: Baseline CPT Class B (12 wk): Includes participants in Cohort B (12 wk) with CPT score B at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort B: Baseline CPT Class B (24 wk): Includes participants in Cohort B (24 wk) with CPT score B at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort B: Baseline CPT Class C (12 wk): Includes participants in Cohort B (12 wk) with CPT score C at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
- Cohort B: Baseline CPT Class C (24 wk): Includes participants in Cohort B (24 wk) with CPT score C at baseline (randomization was based on screening measurement), and who had CPT score assessments at both baseline and Posttreatment Week 4.
Arm/Group | Cohort A: Baseline CPT Class B (12 wk) | Cohort A: Baseline CPT Class B (24 wk) | Cohort A: Baseline CPT Class C (12 wk) | Cohort A: Baseline CPT Class C (24 wk) | Cohort B: Baseline CPT Class A (12 wk) | Cohort B: Baseline CPT Class A (24 wk) | Cohort B: Baseline CPT Class B (12 wk) | Cohort B: Baseline CPT Class B (24 wk) | Cohort B: Baseline CPT Class C (12 wk) | Cohort B: Baseline CPT Class C (24 wk)
Number analyzed (Participants) | 28 | 23 | 17 | 19 | 35 | 34 | 18 | 20 | 2 | 5
percentage of participants
  Decrease | 64.3 | 87.0 | 82.4 | 73.7 | 28.6 | 23.5 | 61.1 | 85.0 | 100.0 | 80.0
  No Change | 28.6 | 13.0 | 11.8 | 26.3 | 68.6 | 61.8 | 33.3 | 10.0 | 0.0 | 20.0
  Increase | 7.1 | 0.0 | 5.9 | 0.0 | 2.9 | 14.7 | 5.6 | 5.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Up to 24 weeks on treatment plus 30 days
Description: Safety Analysis Set: participants who were enrolled and received at least one dose of study drug
Arm/Group | Cohort A, Group 1 (12 wk): CPT Class B (7-9) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis | Cohort B, Group 4 (12 wk): CPT Class A (5-6) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) | Cohort B, Group 7 (12 wk): FCH | Cohort B, Group 7 (24 wk): FCH
Serious Adverse Events (participants affected / at risk) | 3/28 | 6/28 | 13/25 | 10/26 | 9/52 | 5/49 | 3/34 | 7/33 | 5/22 | 6/23 | 1/3 | 2/5 | 2/3 | 1/2
Other Adverse Events (participants affected / at risk) | 25/28 | 25/28 | 23/25 | 23/26 | 49/52 | 48/49 | 27/34 | 30/33 | 20/22 | 20/23 | 3/3 | 5/5 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A, Group 1 (12 wk): CPT Class B (7-9) (N=28) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) (N=28) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) (N=25) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) (N=26) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis (N=52) | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis (N=49) | Cohort B, Group 4 (12 wk): CPT Class A (5-6) (N=34) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) (N=33) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) (N=22) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) (N=23) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) (N=3) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) (N=5) | Cohort B, Group 7 (12 wk): FCH (N=3) | Cohort B, Group 7 (24 wk): FCH (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac septal hypertrophy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricle outflow tract obstruction (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device dislocation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver transplant rejection (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endocarditis staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritoneal tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A, Group 1 (12 wk): CPT Class B (7-9) (N=28) | Cohort A, Group 1 (24 wk): CPT Class B (7-9) (N=28) | Cohort A, Group 2 (12 wk): CPT Class C (10-12) (N=25) | Cohort A, Group 2 (24 wk): CPT Class C (10-12) (N=26) | Cohort B, Group 3 (12 wk): F0-F3 Fibrosis (N=52) | Cohort B, Group 3 (24 wk): F0-F3 Fibrosis (N=49) | Cohort B, Group 4 (12 wk): CPT Class A (5-6) (N=34) | Cohort B, Group 4 (24 wk): CPT Class A (5-6) (N=33) | Cohort B, Group 5 (12 wk): CPT Class B (7-9) (N=22) | Cohort B, Group 5 (24 wk): CPT Class B (7-9) (N=23) | Cohort B, Group 6 (12 wk): CPT Class C (10-12) (N=3) | Cohort B, Group 6 (24 wk): CPT Class C (10-12) (N=5) | Cohort B, Group 7 (12 wk): FCH (N=3) | Cohort B, Group 7 (24 wk): FCH (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 5 | 8 | 21 | 27 | 10 | 15 | 6 | 12 | 1 | 1 | 2 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid cyst (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pterygium (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 3 | 1 | 4 | 5 | 3 | 4 | 1 | 2 | 1 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 3 | 0 | 2 | 4 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 2 | 5 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 3 | 3 | 12 | 11 | 5 | 11 | 2 | 3 | 1 | 2 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 5 | 4 | 1 | 4 | 0 | 2 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 4 | 4 | 5 | 13 | 6 | 5 | 10 | 6 | 3 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 6 | 3 | 5 | 3 | 4 | 4 | 3 | 4 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 2 | 2 | 3 | 4 | 4 | 4 | 5 | 7 | 1 | 4 | 1 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 10 | 9 | 5 | 8 | 22 | 20 | 8 | 11 | 7 | 9 | 1 | 1 | 1 | 1
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 2 | 1 | 7 | 0 | 0 | 3 | 2 | 2 | 2 | 0 | 0 | 1 | 1
Peripheral swelling (General disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 4 | 3 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 2 | 1 | 1 | 2 | 2 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 0 | 4 | 5 | 2 | 5 | 1 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Puncture site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 3 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 4 | 1 | 2 | 5 | 3 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 1 | 5 | 4 | 2 | 3 | 2 | 1 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 5 | 5 | 4 | 2 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 5 | 4 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 1 | 3 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 3 | 1 | 2 | 7 | 5 | 3 | 1 | 2 | 2 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 8 | 7 | 7 | 2 | 12 | 14 | 6 | 9 | 2 | 7 | 0 | 1 | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0
Lethargy (Nervous system disorders) | 2 | 0 | 3 | 3 | 1 | 3 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 4 | 4 | 4 | 8 | 10 | 4 | 3 | 2 | 4 | 1 | 0 | 1 | 1
Irritability (Psychiatric disorders) | 2 | 1 | 1 | 1 | 2 | 3 | 2 | 3 | 0 | 2 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 1 | 1 | 4 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 4 | 4 | 5 | 8 | 4 | 7 | 3 | 4 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3 | 9 | 4 | 5 | 3 | 2 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 5 | 3 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 2 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 8 | 3 | 4 | 5 | 6 | 4 | 7 | 2 | 2 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 2 | 2 | 4 | 3 | 4 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years